CLINICAL TRIAL: NCT03052491
Title: Effects of a Multi-Pathway Dietary Supplement (Stem Cell 100+) on Indices of Health and Life Expectancy
Brief Title: Effects of a 10 Component Dietary Supplement on Health and the Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centagen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SC100+ Clinical #1
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Blood Pressure; HDL Low; Stress; Lung Function Decreased; Quality of Life; Energy Supply; Deficiency; Concentration Ability Impaired; Joint Instability; Immune Deficiency
MeSH Terms: conditions — Respiratory Insufficiency; Joint Instability; Immunologic Deficiency Syndromes

STUDY DESIGN:
Intervention Model Description: Open-label field trial without a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem Cell 100+ Intervention (Experimental): Subjects take one 650 mg capsule by mouth twice daily for an average of 15 weeks
  Interventions: Dietary Supplement: Stem Cell 100+

INTERVENTIONS:
Dietary Supplement: Stem Cell 100+ — Open-Label 10-Component Dietary Supplement
  Other Names: SC100+

SUMMARY:
This open-label field trial evaluates the effects of treatment with a multi-pathway dietary supplement (Stem Cell 100+) that has been commercially available for several years. The objective of the intervention trial is to determine if normal subjects over 35 years of age experience any observable health benefits from the dietary supplement as to their blood pressure, pulse rate, blood cholesterol, lung capacity, stress levels, or self reported changes in markers of overall health and life expectancy.

DETAILED DESCRIPTION:
Currently, only dietary restriction has been verified to slow the rate of aging and to promote general health. This trial is designed to see whether a complex supplement (Stem Cell 100+) that targets multiple longevity pathways could also have positive effects on several markers of successful aging and good health. Multipath causes of aging include: stem cell function, telomere loss, chronic stress, inflammation, insulin-like growth factors, autophagy, vascular loss, neural dysfunction, and oxidative stress. The goal of the study was to test the effects of this novel multipath intervention strategy in a clinical trial of healthy people using health markers such as blood pressure, cholesterol status, lung function, stress levels, and self-reported health status. Hundreds of published animal and human clinical studies have been done with each of the individual active ingredients in the formulation, which target many critical causes of aging.

Based on their published animal studies showing extension of life span in a model animal and their laboratory work on adult human stem cells, the investigators believe that Stem Cell 100+ will provide evidence of efficacy in addressing multiple index markers of health and life expectancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* No history of serious cardiovascular, cancer, or neural disease.
* Normal health for age
* Willing to have blood drawn at baseline and after trial
* Willing to submit to evaluation testing of blood pressure, lung testing, stress testing.
* Willing to take online self reported survey of health at end of trial

Exclusion Criteria:

* History of metastatic cancer, heart attack, dementia, or other life-threatening disease
* Any subject who is not capable of responding to a self-reported online questionnaire
* Pregnant

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03-12 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Baseline and at an average of 15 weeks
  Change in Systolic and Diastolic Blood Pressure
HDL Cholesterol | Baseline and at an average of 15 weeks
  Change in HDL Cholesterol
Lung Capacity | Baseline and at an average of 15 weeks
  Change in Peak Expiatory Flow
Stress Level | Baseline and at an average of 15 weeks
  Change in Heart Rate Variability
Heart Rate | Baseline and at an average of 15 weeks
  Change in Heart Rate

SECONDARY OUTCOMES:
Overall Health | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Ability to Concentrate or Focus | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Joint Flexibility | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Work Productivity | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Ability to Relax | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Cold/Flu Resistance | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Stress Tolerance | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Energy Level | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Endurance | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Ease of Walking | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Climbing Stairs | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Overall Mood | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)
Vitality | From baseline through study completion, an average of 15 weeks
  Self-Reported Change based on a 7 point range from Much Better (+3) to Much Worse (-3)

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Villeponteau, Ph.D., Principal Investigator — Centagen, Inc.
Locations (1):
- Accelagen, Inc., San Diego, California, United States

REFERENCES:
- [Background] Villeponteau B, Matsagas K, Nobles AC, Rizza C, Horwitz M, Benford G, Mockett RJ. Herbal supplement extends life span under some environmental conditions and boosts stress resistance. PLoS One. 2015 Apr 16;10(4):e0119068. doi: 10.1371/journal.pone.0119068. eCollection 2015. PMID 25879540
- [Background] Villeponteau B, Cockrell R, Feng J. Nutraceutical interventions may delay aging and the age-related diseases. Exp Gerontol. 2000 Dec;35(9-10):1405-17. doi: 10.1016/s0531-5565(00)00182-0. PMID 11113618
- [Background] Villeponteau B. The heterochromatin loss model of aging. Exp Gerontol. 1997 Jul-Oct;32(4-5):383-94. doi: 10.1016/s0531-5565(96)00155-6. PMID 9315443
- [Background] Marusic L, Anton M, Tidy A, Wang P, Villeponteau B, Bacchetti S. Reprogramming of telomerase by expression of mutant telomerase RNA template in human cells leads to altered telomeres that correlate with reduced cell viability. Mol Cell Biol. 1997 Nov;17(11):6394-401. doi: 10.1128/MCB.17.11.6394. PMID 9343401
- [Background] Harley CB, Villeponteau B. Telomeres and telomerase in aging and cancer. Curr Opin Genet Dev. 1995 Apr;5(2):249-55. doi: 10.1016/0959-437x(95)80016-6. PMID 7613096
- See also: Wikipedia description of Villeponteau's contributions to science and medicine — http://en.wikipedia.org/wiki/Bryant_Villeponteau